CLINICAL TRIAL: NCT03161119
Title: Prospective Randomized Controlled Trial Comparing Two Different Embryo Transfer (ET) Catheters
Brief Title: Comparing Two Different Embryo Transfer Catheters
Acronym: CATH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1610
Record Dates: First submitted 2017-05-04; First posted 2017-05-19 (Actual); Last update posted 2019-03-21 (Actual); Status verified 2018-06

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Catheter Cook K-Jets-551910-S (Experimental): Catheter Cook K-Jets-551910-S consists of an outer firm and an inner ultrasoft catheter. The outer guiding catheter (17 cm long) is slightly stiff, with a preshaped curve and a rounded bulb tip to help negotiate the cervical canal. It has a depth marker at 4 cm from the tip, which can be pulled back to a second marker at 5 cm. The inner catheter (23 cm long) is made of a soft material with a rounded bullet tip. In general, the inner catheter does not negotiate the cervical canal directly but rather is introduced into the uterine cavity through the outer catheter.
  Interventions: Device: Ultrasound guided embryotransfer with Cook K-Jets-551910-S
- Catheter Cook k-soft-5000 (or K-J-SP-681710, K-J-SPPE-68171) (Active Comparator): This catheter system consists of an outer firm and inner soft catheter. The outer guiding catheter (15,4 cm long) is straight and made of flexible material. The inner catheter (23 cm long) is made of a very soft and flexible polyurethan. The inner catheter is introduced directly through the cervix.
  Interventions: Device: Ultrasound guided embryotransfer with Cook k-soft-5000 (or K-J-SP-681710 and K-J-SPPE-681710)

INTERVENTIONS:
Device: Ultrasound guided embryotransfer with Cook K-Jets-551910-S — On the day of ET, patient will be asked to come with full bladder. ET will be done with patient in lithotomy position. No anesthesia will be used for the procedure. Under sterile condition, vaginal parts will be cleaned with saline and draped and speculum inserted to expose cervix. Cervical mucus and cervix will be cleaned with sterile media.
  The Et procedure itself is standardized as far as possible amongst the participating physicians to eliminate bias.
  Arms: Catheter Cook K-Jets-551910-S
Device: Ultrasound guided embryotransfer with Cook k-soft-5000 (or K-J-SP-681710 and K-J-SPPE-681710) — On the day of ET, patient will be asked to come with full bladder. ET will be done with patient in lithotomy position. No anesthesia will be used for the procedure. Under sterile condition, vaginal parts will be cleaned with saline and draped and speculum inserted to expose cervix. Cervical mucus and cervix will be cleaned with sterile media.
  The Et procedure itself is standardized as far as possible amongst the participating physicians to eliminate bias.
  Arms: Catheter Cook k-soft-5000 (or K-J-SP-681710, K-J-SPPE-68171)

SUMMARY:
Numerous published trials now document that the embryo transfer (ET) procedure has a huge impact on pregnancy and delivery rates after IVF (In Vitro Fertilization).

To compare the ease of use (defined as the rate of successful atraumatic insertion) of different types of embryo transfer (ET) catheters.

This prospective randomized unblinded controlled clinical trial is performed to determine if there is any difference in ease of use among 2 different catheters : Cook k-soft-5000, Cook K-JETS-551910-S.

Inclusion criteria: patients < / = 38 years of age, body mass index (BMI) between 18 and 28, at least one frozen-thawed blastocyst transferred.

Exclusion criteria: ICSI (Intracytoplasmic Sperm Injection)-TESE (Testicular Sperm Extraction) IVF cycles.

A number of 352 consecutive women undergoing embryo transfer will be selected for this prospective, randomized controlled trial. Two protocols for endometrial preparation will be used before frozen/thawed blastocyst transfer: the modified spontaneous protocol and the oral/transdermal preparation protocol. ET will be done with patient in lithotomy position, under ultrasound guidance. No anesthesia will be used for the procedure.

176 patients will be enrolled in this trial and randomized to enter one of the two catheter group.

DETAILED DESCRIPTION:
Introduction

Embryo transfer (ET) is the final and critical step in the long pathway of in vitro fertilization (IVF) treatment. Implantation is a complex process and, as yet, one not fully understood. Aside from the quality of the embryos replaced and the receptivity of the endometrium, the embryo transfer procedure itself might impact the implantation process.

The procedure has changed very little since the first descriptions. Numerous data suggest that difficult transfers should be avoided, as they are likely to reduce the chances of implantation and subsequent pregnancy rates.

It has been proposed on the basis of small studies that traumatic embryo transfer can induce uterine contractions capable of displacing the embryo or induce unwanted endometrial damage. The evidence is unclear, however, as whilst several studies support this concept, others do not.

Free hand embryo transfer with soft catheters under ultrasound guidance is considered the best option in transferring embryos. Many retrospective trials have reported higher Pregnancy Rates (PR) with soft catheters compared with hard catheters. However in technically difficult ET, where difficulties are met in negotiating the cervical os, the use of harder catheters is needed. The change from soft to hard catheters in these transfers, along with the difficulty of the transfer itself, may account for differences in pregnancy rate.

On the other hand it is likely that the experience of the clinicians and their confidence with the catheter are the main variables involved in this 'artistic' skill.

On the basis of a large recent RCT, variations in the PR may depend on variations between operators and their confidence with different type of catheters.

The investigators work in a large teaching hospital where many different operators with different levels of experience perform ET. The rate of difficult ET varies considerably between operators (between 15% and 42%, median 30%) although the overall PR does not vary significantly. With this study the investigators would like to point out whether or not there is a catheter that is able to significantly reduce the difficult transfer rate. The secondary outcome is to assess if one of the catheters is able to sensibly minimize the differences in difficult transfer rate between operators.

Objective

Assessing differences in terms of difficult embryo-transfer rate among two different type of catheter: Cook k-soft-5000 (or K-J-SP-681710 and K-J-SPPE-681710) and Cook K-JETS-551910-S. In order to achieve a measurable difference in the ease of use of the two catheters we decided to compare the median percentage of 'difficult transfer' for all the operators performing the included ETs with the two different catheters. Moreover we aim to study the percentage of difficult ET among operators with the two ET catheters in order to highlight if different catheters may be associated to different interoperator variability in difficult ET rate.

Materials and Methods 352 consecutive women undergoing frozen/thawed blastocyst transfer will be selected for this prospective, randomized controlled trial. The frozen blastocysts result from supernumerary embryos or from 'freeze all policy' in patients at high risk of Severe Ovarian Hyperstimulation Syndrome (OHSS).

The randomization of the single patient to one of the two study branches will be done by the nurse or the embryologist just before the procedure.

Endometrial preparation (modified spontaneous cycle and pharmacological endometrial preparation) Modified Spontaneous cycle In patient with regular menses, the endometrial thickness and dominant follicle diameter are monitored with transvaginal scan beginning on day 8 since period onset. When preovulatory follicle reaches the mean diameter of at least 16 mm a vial of hCG (human Chorionic Gonadotropin) 5000 IU is administered subcutaneously, intravaginal Progesterone is started 2 days later and the blastocyst transfer is scheduled 7 days after hCG injection.

Pharmacological Endometrial preparation In patient with irregular menses, endometrial preparation with oral or transdermal oestradiol is prescribed and started on day 2 of the period. Endometrial thickness and ovarian quiescence are monitored via transvaginal scan starting on day 10-12 since the period onset. When endometrial thickness reaches a minimum of 7,5 mm, intravaginal progesterone is started and blastocyst transfer is performed 5 days later.

Technique of ET On the day of ET, patient will be asked to come with a full bladder. ET will be done with patient in lithotomy position. No anesthesia will be used for the procedure. Under sterile condition, speculum is inserted to expose cervix, cervix will be cleaned with sterile physiologic solution and gently draped.

The Et procedure itself is standardized as far as possible amongst the participating physicians to eliminate bias.

Description of Transfer technique with the two different catheters.

* Catheter Cook K-Jets-551910-S consists of an outer firm and an inner ultrasoft catheter. The outer guiding catheter (17 cm long) is slightly stiff, with a preshaped curve and a rounded bulb tip to help negotiate the cervical canal. It has a depth marker at 4 cm from the tip, which can be pulled back to a second marker at 5 cm. The inner catheter (23 cm long) is made of a soft material with a rounded bullet tip. In general, the inner catheter does not negotiate the cervical canal directly but rather is introduced into the uterine cavity through the outer catheter.
* Catheter Cook k-soft-5000 (or K-J-SP-681710 and K-J-SPPE-681710): this catheter system consists of an outer firm and inner soft catheter. The outer guiding catheter (15,4 cm long) is straight and made of flexible material. The inner catheter (23 cm long) is made of a very soft and flexible polyurethan. The inner catheter is introduced directly through the cervix.

Easy transfers are defined as follows:

* Cook k-soft-5000 catheter: straight-forward advancing of the preloaded inner catheter through the cervix, the internal os and the uterine cavity up to the site of embryo release, chosen on the basis of an acceptable Ultrasound vision.
* Cook K-JETS-551910-S catheter: straight-forward advancement of the outer catheter through the cervix up to the internal os followed by straight-forward advancement of the inner loaded catheter from outer catheter tip to the site of embryo release, chosen on the basis of acceptable Ultrasound vision.

Difficult transfers are defined as follow:

* Cook k-soft-5000 catheter (or K-J-SP-681710 and K-J-SPPE-681710): advancement of the outer sheath, multiple attempts, force, required manipulation, use of a stylet or tenaculum, dilatation;
* Cook K-JETS-551910-S catheter: required manipulation, multiple attempts, force, the use of a stylet or tenaculum, dilatation.

Pregnancy assessment Clinical pregnancy will be defined as follows: a pregnancy diagnosed by ultrasonographic visualization of one or more gestational sacs or definitive clinical signs of pregnancy. It includes ectopic pregnancy. Live birth was defined as delivery of a living baby after at least 24 weeks of gestation.

Numerosity The sample size has been calculated on the basis of historical difficult Et rate registered in years 2014 and 2015.

In the period 01/01/2014-31/12/2015 a total of 1014 ET were performed. We calculated a 28 % of difficult ET with a 30% median of difficult transfer rate among all operators and the number of operators performing the procedure was 22.

In order to detect a 50 % difference in difficult ET rate (90% power), 352 patients need to be enrolled in the study (176 patients per group).

Data Management The data collected on the ET will be registered in a specific database in which each patient will be identified by an identification code.

Patients enrolled in this trial will have consented in writing that their medical records could be used for research purposes, as long as the patients' anonymity was protected and confidentiality of the medical record was assured.

ELIGIBILITY:
Inclusion Criteria:

* body mass index (BMI) between 18 and 28,
* at least one frozen/thawed blastocyst

Exclusion Criteria:

* ICSI-TESE cycles

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 352 (Estimated)
Dates: Start 2017-09-26 (Actual); Primary Completion 2019-06-01 (Estimated); Study Completion 2019-12-01 (Estimated)

PRIMARY OUTCOMES:
Prevalence of difficult transfers (Number of difficult transfers/ Total transfers) | through study completion, 18 months
  Difficult transfers are defined as
  1. for Cook k-soft-5000 catheter: advancement of the outer sheath, multiple attempts, force, required manipulation, use of a stylet or tenaculum, dilatation;
  2. for Cook K-JETS-551910-S catheter: required manipulation, multiple attempts, force, the use of a stylet or tenaculum, dilatation.

SECONDARY OUTCOMES:
Inter-operator variability in prevalence of difficult transfers with the 2 catheters | through study completion, 18 months
  prevalence of difficult transfer rate as defined above and inter operator variability.

CONTACTS AND LOCATIONS:
Overall Officials: Paolo E Levi Setti, Study Director — Istituto Clinico Humanitas
Locations (1):
- Paolo Emanuele Levi Setti, Rozzano, MI, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Levi Setti PE, Cirillo F, Morenghi E, Immediata V, Caccavari V, Baggiani A, Albani E, Patrizio P. One step further: randomised single-centre trial comparing the direct and afterload techniques of embryo transfer. Hum Reprod. 2021 Aug 18;36(9):2484-2492. doi: 10.1093/humrep/deab178. PMID 34323282